CLINICAL TRIAL: NCT06359353
Title: Effect of Pitavastatin on Bone Metabolism in Patients With Hypercholesterolemia and Low Bone Mass
Brief Title: Effect of Pitavastatin on Bone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B-1902-520-004
Record Dates: First submitted 2024-04-01; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Osteoporosis, Osteopenia; Hypercholesterolemia; Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Hypercholesterolemia; Osteoporosis, Postmenopausal | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pitavastatin (Experimental): Pitavastatin 2 mg or 4 mg once daily
  * The dosage is determined based on cholesterol levels and the physician's decision.
  Interventions: Drug: Pitavastatin

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin 2 mg or 4 mg once daily
  * The dosage is determined based on cholesterol levels and the physician's decision.
  Other Names: Livalo tab

SUMMARY:
This clinical trial investigates the effects of pitavastatin on bone health in postmenopausal women with osteopenia or osteoporosis and hypercholesterolemia. Given the high prevalence of osteoporosis in aging populations and the associated risks, even with existing treatments, this study addresses a critical gap in medical research. Statins, specifically HMG-CoA reductase inhibitors, are suggested to benefit bone metabolism by promoting bone formation and reducing resorption. However, the specific impact of pitavastatin on bone metabolism lacks clinical evidence.

The study's primary goal is to determine the effects of a 12-month pitavastatin regimen on bone metabolism markers in this population. This research could significantly contribute to developing more effective osteoporosis treatments for postmenopausal women, combining bone health and cholesterol management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are under the age of 75 and are postmenopausal.
* Individuals diagnosed with osteopenia or osteoporosis, exhibiting a T-score ranging from -3.0 to -1.5.
* Patients with hypercholesterolemia starting pitavastatin for the first time.
* Patients exhibiting baseline bone resorption markers, specifically C-telopeptide levels of 0.300 ng/mL or above, or NTX levels above 16.5 nmolBCE/L.

Exclusion Criteria:

* Patients who have used a statin medication for more than one month within the last 3 months.
* Patients who have used oral or injectable glucocorticoids for more than one week within the last 3 months.
* Patients currently using thiazolidinediones, a class of oral antidiabetic medications.
* Patients undergoing treatment for malignant tumors.

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Change in blood urinary N-Telopeptide of Type I Collagen levels compared to baseline after 6 months | 6 month
  nmol BCE/L

SECONDARY OUTCOMES:
Change in blood C-Telopeptide of Type I Collagen levels | 6 and 12 months
  ng/L
Change in blood Osteocalcin levels | 6 and 12 months
  ng/mL
Change in urinary N-Telopeptide of Type I Collagen levels | 6 and 12 months
  nmol BCE/L
Change in blood Procollagen Type 1 N-Terminal Propeptide levels | 6 and 12 months
  ng/mL
Change in blood LDL-cholesterol levels | 6 and 12 months
  mg/dL
Change in blood HbA1c levels | 6 and 12 months
Changes in bone mineral density | 12 months
  measured by dual-energy X-ray absorptiometry

OTHER OUTCOMES:
Changes of the outcomes after 12 months | 24 months, up to 36 months
  bone mineral density and bone metabolism markers

CONTACTS AND LOCATIONS:
Overall Officials: Soo Soo, M.D. Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided